CLINICAL TRIAL: NCT05505279
Title: Does High Flow Nasal Canula (HFNC) Prevent Hypercapnia During EBUS Under Procedural Sedation?
Brief Title: Ventilatory Effects of THRIVE During EBUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-2031
Record Dates: First submitted 2022-08-10; First posted 2022-08-17 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hypercapnia; Sedation Complication; High Flow Nasal Cannula
Keywords: High Flow Nasal Cannula; Sedation; Dead space ventilation
MeSH Terms: conditions — Hypercapnia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient is sedated and the investigators are blinded for the randomization. Only the care provider is aware of the randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30 L - 70 L (Active Comparator): Initially, all patients will receive 3L/min of oxygen for 10 minutes. Than, patients in this arm will receive 30L/min of High Flow Nasal Oxygen for 15 minutes and subsequently 70 L/min for another 15 minutes.
  Interventions: Device: THRIVE (High Flow Nasal Cannula)
- 70 L - 30 L (Active Comparator): Initially, all patients will receive 3L/min of oxygen for 10 minutes. Than, patients in this arm will receive 70L/min of High Flow Nasal Oxygen for 15 minutes and subsequently 30 L/min for another 15 minutes.
  Interventions: Device: THRIVE (High Flow Nasal Cannula)

INTERVENTIONS:
Device: THRIVE (High Flow Nasal Cannula) — 2 different rates of nasal flow compared to each other and a baseline of level of nasal oxygen
  Other Names: THRIVE; Optiflow; High Flow Nasal Cannula; High Flow Nasal Oxygen

SUMMARY:
High flow nasal cannula (HFNC) is used in interventional procedures to prevent hypoxia during sedation. In patients with a patent airway, HFNC reduces dead space ventilation as well. It is unknown if dead space ventilation is also reduced by HFNC in an EndoBroncheal UltraSound procedure, in which the airway is partially blocked by the endoscope. Especially in patients with Chronic Obstructive Pulmonary Disease (COPD) the partial blocking of the airway may reduce ventilation. If HFNC is able to reduce dead space during an EBUS-procedure, it may facilitate CO2 clearance, which may lead to a reduction in work of breathing.

This study aims to investigate if HFNC reduces dead space ventilation in patients undergoing an EBUS-procedure and if this is flow-dependent.

A randomized, double-blinded, cross-over study is designed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COPD Gold classification 3 or 4
* Scheduled EBUS with sedation

Exclusion Criteria:

* Known neurodegenerative diseases, such as Amyotrophic Lateral Sclerosis, dementia, Multiple Sclerosis or Guillain-Barré.
* Allergy or intolerance for propofol or esketamine
* Severe pulmonary hypertension (PAPsyst > 60 mmHg)
* Pregnancy
* upper airway obstruction, such as subglottic stenosis or obstructing tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Inspiratory CO2 at 10 minutes (baseline) | at t=10 minutes
  Inspiratory CO2, measured at the carinal level
Inspiratory CO2 at 25 minutes | at=25 minutes
  Inspiratory CO2, measured at the carinal level
Inspiratory CO2 at 45 minutes | at t=45 minutes
  Inspiratory CO2, measured at the carinal level
expiratory CO2 at 10 minutes (baseline) | at t=10 minutes
  Expiratory CO2, measured at the carinal level
expiratory CO2 at 25 minutes | at t=25 minutes
  Expiratory CO2, measured at the carinal level
expiratory CO2 at 45 minutes | t=45 minutes
  Expiratory CO2, measured at the carinal level
Slope of capnography at 10 minutes (baseline) | At t=10 minutes
  Angle of the D-E segment (inspiratory slope)
Slope of capnography at 25 minutes | At t=25 minutes
  Angle of the D-E segment (inspiratory slope)
Slope of capnography at 45 minutes | At t=45 minutes
  Angle of the D-E segment (inspiratory slope)

SECONDARY OUTCOMES:
Respiratory rate | At t=10 minutes
  Respiratory rate, measured by capnography
Respiratory rate | At t=25 minutes
  Respiratory rate, measured by capnography
Respiratory rate | At t=45 minutes
  Respiratory rate, measured by capnography
The level of HFNC dead space washout | At t=10 minutes
  Levels of inspiratory and expiratory CO2 measured at the level of the left main bronchus, level of carina and the subglottic level.
The level of HFNC dead space washout | At t=25 minutes
  Levels of inspiratory and expiratory CO2 measured at the level of the left main bronchus, level of carina and the subglottic level.
The level of HFNC dead space washout | At t=45 minutes
  Levels of inspiratory and expiratory CO2 measured at the level of the left main bronchus, level of carina and the subglottic level.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miechels, Principal Investigator — Dept. of Anesthesiology and Critical Care, Rijnstate Hospital, Arnhem; Mark V Koning, MD, PhD, Study Chair — Dept. of Anesthesiology and Critical Care, Rijnstate Hospital, Arnhem; Niels Claessens, MD, PhD, Study Director — Dept. of Pulmonology, Rijnstate Hospital, Arnhem
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request and within the limits of the law on patient data distribution.